CLINICAL TRIAL: NCT04087941
Title: Hepatocyte Growth Factor for Opioid-Dependent Pain: Efficacy and Safety of VM202 in Painful Diabetic Peripheral Neuropathy (The HOPES Trial)
Brief Title: Efficacy and Safety of VM202 in Painful Diabetic Peripheral Neuropathy -The HOPES Trial
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: This study never left the planning stages: there was no IRB application and no participants were enrolled.
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Christine N. Sang, MD, MPH, Director, Translational Pain Research, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HOPES
Record Dates: First submitted 2019-09-11; First posted 2019-09-12 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Painful Diabetic Neuropathy
MeSH Terms: conditions — Diabetic Neuropathies

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Biological: VM-202
- VM-202 (Experimental)
  Interventions: Biological: VM-202

INTERVENTIONS:
Biological: VM-202 — VM202 is a DNA plasmid that contains novel genomic cDNA hybrid human hepatocyte growth factor (HGF) coding sequence (HGF-X7) expressing two isoforms of HGF, HGF 728 and HGF 723.

SUMMARY:
A double-blind, randomized, placebo-controlled, single-center, 12-month phase 2 study designed to assess the safety and efficacy of VM202 as a replacement for opioid analgesics in opioid-tolerant subjects with painful diabetic peripheral neuropathy (DPN).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years to 75 years;
2. Documented history of Type I or II diabetes with current treatment control(glycosylated hemoglobin A1c of ≤ 10.0% at Screening) and currently on oral medication and / or insulin;
3. Taking 60 to 200 mg morphine milligram equivalents (MME)/day for painful DPN at study entry and must be on stable regimen starting at Day -21; percent of overall requirement as immediate release must be ≥ 30%;
4. No significant changes anticipated in diabetes medication regimen;
5. No new symptoms associated with diabetes within the last 3 months prior to study entry;
6. Diagnosis of painful diabetic peripheral neuropathy in both lower extremities;
7. Global pain intensity [Numerical rating scale, average NRS] score over the week prior to initial Screening visit must be ≥ 4 and ≤ 9 (0 = no pain - 10 = worst pain imaginable);
8. Symptoms from the Brief Pain Neuropathy Screening (BPNS) is ≤ 5 point difference between legs at Initial Screening;
9. The physical examination component of the Michigan Neuropathy Screening Instrument Score (MNSI) is ≥ 3 at Initial Screening;
10. Subjects on gabapentin (Neurontin), pregabalin (Lyrica), or duloxetine (Cymbalta) for painful DPN at study entry must be on a stable regimen of these treatments for at least 7 days prior to start of oral placebo run-in; and
11. If female of childbearing potential, negative urine pregnancy test at screening and using acceptable method of birth control during the study.

Exclusion Criteria:

1. Small fiber polyneuropathy caused by condition other than diabetes;
2. Additional pain syndrome of overall greater intensity than that of DPN that, in the opinion of the investigator, would prevent assessment of DPN;
3. Progressive or degenerative neurological disorder;
4. Myopathy;
5. Inflammatory disorder of the blood vessels (inflammatory angiopathy, such as Buerger's disease);
6. Active infection, in the opinion of the investigator;
7. Chronic inflammatory disease (e.g., Crohn's disease, rheumatoid arthritis), in the opinion of the investigator;
8. Positive HIV or HTLV at Screening;
9. Active Hepatitis B or C as determined by Hepatitis B core antibody (HBcAb; IgG and IgM), antibody to Hepatitis B surface antigen (HBsAb), Hepatitis B surface antigen (HBsAg) and Hepatitis C antibodies (Anti-HCV) at Screening;
10. Subjects with known immunosuppression or currently receiving immunosuppressive drugs, chemotherapy or radiation therapy;
11. Stroke or myocardial infarction within last 3 months;
12. Specific laboratory values at Screening including: Hemoglobin < 8.0 g/dL, WBC < 3,000 cells per microliter, platelet count <75,000/mm3, Creatinine > 2.0 mg/dL; AST and/or ALT > 3 times the upper limit of normal or any other clinically significant lab abnormality which in the opinion of the investigator should be exclusionary;
13. Proliferative retinopathy within 5 years of signing consent or any ophthalmological condition which, in the opinion of the investigator, should be exclusionary; any condition that precludes standard ophthalmologic examination;
14. Uncontrolled hypertension defined as sustained systolic blood pressure (SBP) > 200 mmHg or diastolic BP (DBP) > 110 mmHg at Screening;
15. Subjects with a recent history (< 5 years) of or new screening finding of malignant neoplasm except basal cell carcinoma or squamous cell carcinoma of the skin (if excised and no evidence of recurrence for one year); subjects with family history of colon cancer in any first degree relative are excluded unless they have undergone a colonoscopy in the last 12 months with negative findings;
16. Use of the following drugs / therapeutics is PROHIBITED past Day -14:

    * skeletal muscle relaxants, benzodiazepines (except for stable bedtime dose),
    * capsaicin, local anesthetic creams and patches, isosorbide dinitrate (ISDN) spray,
    * transcutaneous electrical nerve stimulation (TENS), acupuncture
17. If not using gabapentin (Neurontin), pregabalin (Lyrica), duloxetine (Cymbalta), any antidepressants (e.g., amitriptyline and venlafaxine), any other antiepileptics (e.g., valproic acid, carbamazepine, or vigabatrin), subjects must agree not to start these drugs until after Day 180. Subjects on these medications on day of informed consent must maintain a stable dose starting at Day -21 until Day 180; any changes in analgesic regimen after Day 180 are at the discretion of the investigator;
18. Use of certain COX-1/COX-2 inhibitor drug(s), steroids (except inhaled, ocular, or intra-articular steroids), and anti-Vascular Endothelial Growth Factor (VEGF) agents; subjects may be enrolled if willing/able to undergo medication wash-out prior to the first dosing and to refrain from taking these drugs for the duration of the study;
19. Major psychiatric disorder within last 6 months that would interfere with study participation;
20. Body mass index (BMI) > 45 kg/m2 at Screening;
21. Any prior or lower extremity amputation due to diabetic complications;
22. History of illicit drug or alcohol abuse / dependence in the past 2 years, including but not limited to, cocaine, amphetamines, non-prescribed opioids, and non-prescribed benzodiazepines);
23. Use of an investigational drug or treatment in past 6 months; and
24. Unable or unwilling to give informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-11 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Change in 24-hour Morphine Milligram Equivalents (MME) | baseline week to week prior to Day 180
  The percent change in 24-hour MME use from baseline week to the week prior to Day 180 obtained from the Daily Pain and Sleep Interference Diary

SECONDARY OUTCOMES:
Opioid use - mean dose | Day 90, Day 180, Day 270, Day 365
  mean dose of opioid reported in 24-hour MME at each timepoint
Opioid use - percent change from baseline | Day 90, Day 180, Day 270, Day 365
  percent change from baseline in 24-hour MME during the week prior to each timepoint
Opioid use - percent of subjects who are dose-reduced/opioid free | Day 90, Day 180, Day 270, Day 365
  percent of subjects whose daily opioid consumption is reduced by 50% and 100% (opioid-free) at each timepoint
Opioid-Related AE - Cognition | Day 90, Day 180, Day 270, Day 365
  Cognition as measured with Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) assessed at each timepoint
Opioid-Related AE - Bowel Function | Day 90, Day 180, Day 270, Day 365
  Bowel Function Inventory-revised (BFI-R) assessed at each timepoint
Opioid-Related AE - Numerical Opioid Side Effect (NOSE) | Day 90, Day 180, Day 270, Day 365
  NOSE assessed at each timepoint
Efficacy- Change in Average Pain Intensity | baseline week to week prior to Day 180
  the change in average pain intensity from baseline week to the week prior to Day 180 obtained from the daily eDiaries

CONTACTS AND LOCATIONS:
Overall Officials: Christine N. Sang, MD, MPH, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Translational Pain Research, Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No